CLINICAL TRIAL: NCT04952779
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Regulatory Post Marketing Surveillance (rPMS) Study of Xultophy® (Insulin Degludec / Liraglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Brief Title: Regulatory Post Marketing Surveillance (rPMS) Study of Xultophy® (Insulin Degludec/Liraglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4445; 1111-1211-7084 (Other: World Health Organization)
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Xultophy; insulin degludec; Liraglutide; IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xultophy®: Korean adults with type 2 diabetes mellitus (T2DM) initiating Xultophy® under routine clinical practice and according to approved label in Korea.
  Interventions: Drug: Xultophy® (insulin degludec/liraglutide)

INTERVENTIONS:
Drug: Xultophy® (insulin degludec/liraglutide) — Xultophy® is a fixed ratio combination of the long-acting basal insulin, insulin degludec, and the glucagon-like peptide 1 receptor agonist (GLP-1 RA), liraglutide, administered under the skin.
  Patients will be treated according to routine clinical practice at the discretion of the treating physician according to the label approved by MFDS.
  The assignment of the patient to Xultophy® is not decided in advance by the protocol but falls within current practice and the prescription of Xultophy® is clearly separated from the decision to include the patient in the study.
  Other Names: insulin degludec/liraglutide

SUMMARY:
The aim of this study is to assess the safety and effectiveness of Xultophy® initiated according to label in adults with type 2 diabetes mellitus (T2DM) under routine clinical practice conditions. Participants will get Xultophy® as prescribed to them by the study doctor. The study will last for about 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The decision to initiate treatment with commercially available Xultophy® has been made by the participant/Legally Acceptable Representative (LAR) and the study doctor before and independently from the decision to include the participant in this study.
* Informed consent obtained before any study related activities. Study related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age 19 years or older at the time of signing informed consent form.
* Participants diagnosed (clinically) with T2DM and who is scheduled to start treatment with Xultophy® based on the clinical judgment of their treating physician as specified in the approved Korean-Prescribing information (local label).

Exclusion Criteria:

* Participants who are or have previously been on Xultophy® therapy.
* Known or suspected hypersensitivity to Xultophy® (the active substance or any of the excipients).
* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Korean adults with type 2 diabetes mellitus (T2DM) initiating Xultophy® under routine clinical practice and according to approved label in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) by preferred term | baseline (Visit1, 0 week) to 26 weeks
  Count of events

SECONDARY OUTCOMES:
Level 3 hypoglycaemia (severe) or level 2 hypoglycaemia | Visit1 (0 week) to 26 weeks
  Plasma Glucose (PG) less than 54 mg/dL (3.0 mmol/L)
Change in body weight | Visit 1 (0 week), Visit 3 (13 weeks)
  Kilograms
Change in body weight | Visit 1 (0 week), Visit 4 (26 weeks)
  kilograms
Change of Xultophy® dose | Visit 1 (0 week), 13 weeks (Visit 3)
  Units
Change of Xultophy® dose | Visit (0 week), Visit 4 (26 weeks)
  Units
Change in Glycosylated Haemoglobin (HbA1c) | Visit 1 (0 week), Visit 3 (13 weeks)
  Percentage
Change in HbA1c | Visit 1 (0 week), Visit 4 (26 weeks)
  Percentage
Individuals achieving HbA1c target less than 7.0 % | Visit 1 (0 week), Visit 3 (13 weeks)
  Percentage
Individuals achieving HbA1c target less than 7.0 % | Visit 1 (0 week), Visit 4 (26 weeks)
  Percentage
Change in Fasting Blood Glucose/Plasma Glucose (FBG/FPG) | Visit 1 (0 week), Visit 3 (13 weeks)
  mg/dl
Change in Fasting Blood Glucose/Plasma Glucose (FBG/FPG) | Visit 1 (0 week), Visit 4 (26 weeks)
  mg/dl
Change in Post Prandial Blood/Plasma Glucose (PPBG/PPPG) | Visit 1 (0 week), Visit 3 (13 weeks)
  mg/dl
Change in Post Prandial Blood/Plasma Glucose (PPBG/PPPG) | Visit 1 (0 week), Visit 3 (26 weeks)
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 1452, Study Director — Novo Nordisk A/S
Locations (32):
- South Korea (32):
  - Daejeon Endo Internal Medicine Clinic, Daejeon, Cheongsa-ro, Seo-gu
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Isam Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Eulji University Hospital_Daejeon, Daejeon
  - Daejeon Endo Internal Medicine Clinic, Daejeon
  - Chungbuk National University Hospital, Daejeon
  - Dongguk University Ilsan Hospital, Goyang
  - Hyewon Medical Foundation Sejong General Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Dongtan Jeil Women's Hospital, Gyeonggi-do
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Inha University Hospital, Incheon
  - Hanil General Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Sahm Yook Medical Center, Seoul
  - Yonsei Leehyunchul Internal Medicine, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul
  - KangNam Sacred Heart Hospital, Seoul
  - Jae Clinic, Seoul
  - Uijeongbu Eulji university Hospital, Uijeongbu-si
  - Ulsan Hospital, Ulsan
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com